CLINICAL TRIAL: NCT04537156
Title: A Multicenter, Randomized, Double-Blind, Controlled (Bivalent Human Papillomavirus Vaccine (16,18 Type)(E. Coli)) Phase III Clinical Trial to Estimate Efficacy, Immunogenicity and Safty of the Recombinant Human Papillomavirus Vaccine (6,11,16,18,31,33,45,52,58 Type) (E.Coli) in Healthy Women Aged 18 to 45 Years
Brief Title: Efficacy, Immunogenicity and Safety Study of Recombinant Human Papillomavirus Vaccine(6,11,16,18,31,33,45,52,58 Type)(E.Coli)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Xiamen University (Other)
Collaborators: Xiamen Innovax Biotech Co., Ltd (Industry); Beijing Wantai Biological Pharmacy Enterprise Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jun Zhang, professor, Xiamen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HPV-PRO-009
Record Dates: First submitted 2020-08-19; First posted 2020-09-03 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-02

CONDITIONS: Cervical Intraepithelial Neoplasia; Cervical Cancer; Condylomata Acuminata
Keywords: human papillomavirus vaccine; cervical cancer; cervical intraepithelial neoplasia; condylomata acuminata
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms; Condylomata Acuminata | interventions — human papillomavirus vaccine, L1 type 16, 18

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HPV vaccine (6,11,16,18,31,33,45,52,58 Types) (Experimental): Participants in this arm would receive 270μg/0.5ml HPV vaccines (6,11,16,18,31,33,45,52,58 Types).
  Interventions: Biological: Nonavalent HPV vaccine
- HPV vaccine (16,18 Types) (Active Comparator): Participants in this arm would receive 60μg/0.5ml HPV vaccines (16,18 Types).
  Interventions: Biological: Bivalent HPV vaccine

INTERVENTIONS:
Biological: Nonavalent HPV vaccine — Nonavalent HPV vaccine (270μg/0.5ml) administered intramuscularly according to a 0, 1, 6 month vaccination schedule.
  Arms: HPV vaccine (6,11,16,18,31,33,45,52,58 Types)
Biological: Bivalent HPV vaccine — Bivalent HPV vaccine (60μg/0.5ml) administered intramuscularly according to a 0, 1, 6 month vaccination schedule.
  Arms: HPV vaccine (16,18 Types)

SUMMARY:
This phase III clinical study was designed to evaluate the efficacy,immunogenicity and safety of Recombinant Human Papillomavirus Vaccine (6,11,16,18,31,33,45,52,58 Type)(E.Coli) manufactured by Xiamen Innovax Biotech CO., LTD., in healthy women aged 18-45 years old.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged between 18 and 45 years at the first vaccination;
2. Be able to understand and comply with the request of the protocol(e.g. biological specimen collection, diary card entry and attend regular follow-up), and sign written informed consent;
3. Women who agree to use effective contraception within 8 months after the first vaccination, or women who have undergone tubal ligation, benign subtotal hysterectomy, benign ovarian tumor removal, or postmenopausal women;
4. The number of sexual partners so far less than four;
5. Have intact cervix and have no history of physical or surgical treatment;
6. No previous history of sexually transmitted diseases (including syphilis, gonorrhea, chancroid, venereal lymphogranuloma, groin granuloma, etc.);
7. No previous history of abnormal cervical screening results or cervical intraepithelial neoplasia (CIN), and no abnormality in gynecological examination;
8. Sexual intercourse has occurred.

Exclusion Criteria:

1. Participants with acute cervicitis and acute lower genital tract infection, or with obvious condyloma;
2. Participants during menstruation, or have vaginal medication, sexual behavior (including anal, vaginal or external genital contact, regardless of the sex of parterner) within two days (48 hours) before the visit, which may affect gynecological examinations and specimens collection.
3. Axillary temperature > 37.0℃;
4. Participants who have positive urine pregnancy test, or are pregnant or breastfeeding;
5. Have used other investigational or unregistered products (drugs or vaccines) within 30 days before receiving the research vaccine or have participated in another clinical research in the past two years, or plan to use other research or unregistered products or participate in other research during the research period;
6. Long-term use (more than 14 continuous days) of immunosuppressors and other Immunoregulatory agents or systemic corticosteroids (Except intranasal steroid, the use of low dose topical, ophthalmic and inhaled steroid preparations will be permitted.) 6 months prior to vaccination.
7. Administration of immunoglobulin and/or blood products 3 months prior to vaccination or intending to use them during the study.
8. Administration of inactivated vaccine within 14 days before vaccination or live vaccine within 21 days;
9. Fever (Axillary temperature >38.0℃) 3 days prior to vaccination or system administration of antibiotics or antiviral agents (Anti-flu agents include but are not limited to Tamiflu, Tamiflu, Symmetrel and Flumadine) 5 days prior to vaccination.
10. Have received other HPV vaccines or participated in clinical research related to HPV or cervical cancer previously;
11. Immunodeficiency disease, primary disease of important viscera, cancer and autoimmune disease (including systemic lupus erythematosus, rheumatoid arthritis, asplenia or splenectomy due to any condition, and other autoimmune diseases that investigators believe may influence the immune response).
12. History of severe allergy (e.g., anaphylaxis, generalized urticaria, dyspnea, angioedema, and other significant reaction) to any previous vaccines, or allergy to any of the components of investigational vaccine.
13. Asthma, which has been unstable for the past two years and requires emergency treatment, hospitalization, oral or intravenous corticosteroids;
14. Suffered from a serious medical illness;
15. Self-report past coagulation disorders or abnormal coagulation function;
16. Epilepsy, excluding febrile epilepsy under 2 years of age, alcoholic epilepsy 3 years prior to abstinence or simple epilepsy that did not require treatment in the past 3 years;
17. According to the judgement of investigator, various medical, psychological, social, vocational or other factors that are not suitable for participating in the clinical trial.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9327 (Actual)
Dates: Start 2020-09-05 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority of anti-HPV 16 and 18 seroconversion rates and geometric mean concentrations at Months 7 (type specific neutralizing antibody) in the PPS-I set | Specific neutralizing antibodies at 7 months after first dose
  Detect the level of anti-HPV 16 and 18 specific neutralizing antibodies at one month after the third dose to determine whether nine-valent HPV vaccine is non-inferior to the control bivalent HPV vaccine
Persistent infection of HPV31, 33, 45, 52 and 58 (over 12 months) (Combined analysis of the 5 types) in the mITT-PI set | Cumulative incidence of this endpoint events in 78 months after the first dose
  To evaluate the efficacy of the nine-valent vaccine against this outcome compared with the control vaccine
Incidence of CIN2 + and/or VIN2 + and/or VaIN2 + lesions related to HPV 31, 33, 45, 52 or 58 (Combined analysis of the 5 types) in the mITT-E when the first two endpoints are satisfied | Cumulative incidence of this endpoint events in 78 months after the first dose
  To evaluate the efficacy of the nine-valent vaccine against this outcome compared with the control vaccine

SECONDARY OUTCOMES:
Efficacy1: Incidence of CIN2 + and/or VIN2 + and/or VaIN2 + lesions related to HPV 31, 33, 45, 52 or 58(Combined analysis of the 5 types) and genital warts related to HPV 6, 11 (Combined analysis of each type) | Cumulative incidence of this endpoint events in 78 months after the first dose
  To evaluate the efficacy of the nine-valent vaccine against this outcome compared with the control vaccine
Efficacy2: Incidence of CIN1 + and/or VIN1 + and/or VaIN1 + lesions related to HPV 31, 33, 45, 52 or 58(Combined analysis of the 5 types) and genital warts related to HPV 6, 11 (Combined analysis of each type) | Cumulative incidence of this endpoint events in 78 months after the first dose
  To evaluate the efficacy of the nine-valent vaccine against this outcome compared with the control vaccine
Efficacy3: Incidence of Persistent infection of HPV31, 33, 45, 52 and 58 (transient infection and over 6 months) (Combined analysis of the 5 types) | Cumulative incidence of this endpoint events in 78 months after the first dose
  To evaluate the efficacy of the nine-valent vaccine against this outcome compared with the control vaccine
Efficacy4: Incidence of CIN1 + and/or VIN1 + and/or VaIN1 + lesions related to HPV 31, 33, 45, 52 or 58(Combined analysis of the 5 types) | Cumulative incidence of this endpoint events in 78 months after the first dose
  To evaluate the efficacy of the nine-valent vaccine against this outcome compared with the control vaccine
Efficacy5: Incidence of Persistent infection of HPV31, 33, 45, 52 and 58 (over 6 months) and/or incidence of CIN1 + and/or VIN1 + and/or VaIN1 + lesions related to HPV 31, 33, 45, 52 or 58(Combined analysis of the 5 types) | Cumulative incidence of this endpoint events in 78 months after the first dose
  To evaluate the efficacy of the nine-valent vaccine against this outcome compared with the control vaccine
Efficacy6: Incidence of genital warts related to HPV 6, 11 | Cumulative incidence of this endpoint events in 78 months after the first dose
  To evaluate the efficacy of the nine-valent vaccine against this outcome compared with the control vaccine
Efficacy7: Incidence of Persistent infection of HPV31, 33, 45, 52, 58, 6 and 11 (transient infection and over 6 months and over 12 months) (Combined analysis of the 7 types) | Cumulative incidence of this endpoint events in 78 months after the first dose
  To evaluate the efficacy of the nine-valent vaccine against this outcome compared with the control vaccine
Efficacy8: Incidence of Persistent infection of HPV31, 33, 45, 52, 58, 6 and 11 (over 6 months and over 12 months) (Independent analysis of each type) | Cumulative incidence of this endpoint events in 78 months after the first dose
  To evaluate the efficacy of the nine-valent vaccine against this outcome compared with the control vaccine
Immunogenicity1: Anti-HPV 6, 11, 16, 18, 31, 33, 45, 52, and 58 seroconversion rates and geometric mean concentrations at Months 7 | Month 7 after first vaccination
  Analysis the seroconversion and geometric mean concertration of the type specific antibodies of the 7 types.
Immunogenicity2: Anti-HPV 6, 11, 16, 18, 31, 33, 45, 52, and 58 seroconversion rates and geometric mean concentrations at Months 18 and 30 | Month 18 and 30 after first vaccination
  Analysis the seroconversion and geometric mean concertration of the type specific antibodies of the 7 types.
Immunogenicity3: Anti-HPV 6, 11, 16, 18, 31, 33, 45, 52, and 58 seroconversion rates and geometric mean concentrations at Months 42, 54, 66 and 78 | Month 42, 54, 66 and 78 after first vaccination
  Analysis the seroconversion and geometric mean concertration of the type specific antibodies of the 7 types.
Safety1: Local and systematic adverse events/reactions occurred within 7 days after each vaccination | During the 7-day (Day 0-6) period following each vaccination
  safety analysis
Safety2: Adverse events/reactions occurred within 30 days after each vaccination | Within 30 days (Day 0-30) after any vaccination
  safety analysis
Safety3: Serious adverse events occurred throughout the study | Up to 78 month
  safety analysis. To evaluate number of SAEs compared with the control vaccine.
Safety4: Pregnancy and pregnancy outcome | Up to 78 month
  safety analysis. To evaluate number of births and terminations compared with the control vaccine.
Safety5: New-onset acute and chronic diseases (especially autoimmune diseases) | Up to 78 month
  safety analysis.To evaluate number of new-onset acute and chronic diseases (especially new-onset autoimmune diseases) throughout the study.

OTHER OUTCOMES:
Incidence of CIN2 + and/or VIN2 + and/or VaIN2 + lesions related to HPV 16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59 or 68 (Combined analysis of the high risk types) | Cumulative incidence of this endpoint events in 78 months after the first dose
  To evaluate the efficacy of the nine-valent vaccine against this outcome compared with the control vaccine
Incidence of CIN1 + and/or VIN1 + and/or VaIN1 + lesions related to HPV 16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59 or 68 (Combined analysis of the high risk types) | Cumulative incidence of this endpoint events in 78 months after the first dose
  To evaluate the efficacy of the nine-valent vaccine against this outcome compared with the control vaccine
Incidence of Persistent infection of HPV35, 39,51,56,59 and 68 (total infection and over 6 months and over 12 months) (Independent analysis of each type) | Cumulative incidence of this endpoint events in 78 months after the first dose
  To evaluate the efficacy of the nine-valent vaccine against this outcome compared with the control vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, master, Study Chair — Xiamen University; Hong-xing Pan, master, Principal Investigator — Jiangsu Provincial Centre for Disease Control and Prevention
Locations (2):
- China (2):
  - Jiangsu Provincial Centre for Disease Control and Prevention, Nanjing, Jiangsu
  - Sichuan Provincial Centre for Disease Control and Prevention, Chengdu, Sichuan